CLINICAL TRIAL: NCT03283410
Title: Determination of Propofol Target Concentration for Young and Elderly by Suppression Rate Analysis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Local problems with BIS monitor, we wont have it anymore.
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Head of Anesthesiology, Brasilia University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CAEE 41471115.1.0000.5558
Record Dates: First submitted 2015-05-29; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Anesthesia
Keywords: propofol; dose-response; elderly; young adults
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Study Arm (Experimental): All patients will be sequentially allocated in the single study arm. All patients will receive some propofol dose.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol plasmatic concentration (Marsh)
  Other Names: Diprivan

SUMMARY:
Propofol's dose-response curve is know for the average adult but propofol's plasmatic concentration under total intravenous anesthesia differences between young and elderly must be modeled. Adaptative clinical trial (Dixon's Up and Down) for determination of ED95% of propofol concentration for hypnosis under general anesthesia for young and elderly adults.

DETAILED DESCRIPTION:
Propofol's dose-response curve is know for the average adult but propofol's plasmatic concentration under total intravenous anesthesia differences between young and elderly must be modeled. Method: adaptative clinical trial (Dixon's Up and Down method) for determination of ED95% of propofol concentration (plasmatic, Marsh model) for hypnosis (BIS ranging from 40 to 60) under general anesthesia for young and elderly adults.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Between 18-28 or 65-75 years old
* ASA physical status I or II
* no pre-anesthetic medications prescribed
* scheduled for surgery under general anesthesia
* willing to participate and sign informed consent.

Exclusion Criteria:

* Contraindications for propofol usage
* history of neurologic or psychiatric diseases
* drug abusers
* users of drugs that alter central nervous system
* pregnancy
* emergency surgeries
* rapid sequence intubation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
BIS value greater than 60 or lower than 40 during general anesthesia | BIS value greater than 60 or lower than 40 during general anesthesia
  BIS value greater than 60 or lower than 40 during general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimaraes, MsC, Principal Investigator — Professor